CLINICAL TRIAL: NCT00877006
Title: An Open-Label, Randomized, Parallel-Group Study of Bendamustine Hydrochloride and Rituximab (BR) Compared With Rituximab, Cyclophosphamide, Vincristine, and Prednisone (R-CVP) or Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone (R-CHOP) in the First-Line Treatment of Patients With Advanced Indolent Non-Hodgkin's Lymphoma (NHL) or Mantle Cell Lymphoma (MCL)
Brief Title: Study of Bendamustine Hydrochloride and Rituximab (BR) Compared With R-CVP or R-CHOP in the First-Line Treatment of Patients With Advanced Indolent Non-Hodgkin's Lymphoma (NHL) or Mantle Cell Lymphoma (MCL) - Referred to as the BRIGHT Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C18083/3064/NL/MN
Record Dates: First submitted 2009-04-03; First posted 2009-04-07 (Estimated); Results first posted 2014-04-28 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Non-Hodgkin's Lymphoma; Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Mantle-Cell | interventions — Bendamustine Hydrochloride; Rituximab; Vincristine; Prednisone; Cyclophosphamide; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bendamustine and Rituximab (BR) (Experimental): Participants received the investigational bendamustine and rituximab regimen for 6 to 8 28-day cycles: bendamustine 90 mg/m^2 intravenous (IV) on Days 1 and 2; rituximab 375 mg/m^2 IV on Day 1
  Interventions: Drug: bendamustine; Drug: rituximab
- R-CHOP/R-CVP (Active Comparator): Participants received the standard regimen (R-CHOP or R-CVP) for 6 to 8 21-days cycles.
  R-CHOP: rituximab 375 mg/m^2 IV on Day 1; vincristine 1.4 mg/m^2 (up to 2 mg/m^2 maximum dose) IV on Day 1; doxorubicin 50 mg/m^2 IV Day 1; cyclophosphamide 750 mg/m^2 IV Day 1; prednisone 100 mg oral on Days 1 to 5
  R-CVP: rituximab 375 mg/m^2 IV on Day 1; cyclophosphamide 750 mg/m^2 IV on Day 1 or cyclophosphamide 1000 mg/m^2 IV on Day 1; vincristine 1.4 mg/m^2 (up to 2 mg/m^2 maximum dose) IV on Day 1; prednisone 100 mg oral on Days 1 to 5
  Interventions: Drug: rituximab; Drug: vincristine; Drug: prednisone; Drug: cyclophosphamide; Drug: doxorubicin

INTERVENTIONS:
Drug: bendamustine
  Other Names: Treakisym; Ribomustin; Levact; Treanda; SDX-105
  Arms: Bendamustine and Rituximab (BR)
Drug: rituximab
  Other Names: Rituxan; MabThera; Zytux
Drug: vincristine
  Other Names: Oncovin
  Arms: R-CHOP/R-CVP
Drug: prednisone
  Arms: R-CHOP/R-CVP
Drug: cyclophosphamide
  Other Names: Endoxan; Cytoxan; Neosar; Procytox; Revimmune
  Arms: R-CHOP/R-CVP
Drug: doxorubicin
  Other Names: Adriamycin
  Arms: R-CHOP/R-CVP

SUMMARY:
The primary objective of the study is to compare the complete response (CR) rate of bendamustine and rituximab (BR) with that of standard treatment regimens of either rituximab, cyclophosphamide, vincristine, and prednisone (R-CVP) or rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone (R-CHOP) in patients with advanced, indolent non-Hodgkin's lymphoma (NHL) or mantle cell lymphoma (MCL).

ELIGIBILITY:
Key Inclusion Criteria:

* Histopathologic confirmation of one of the following cluster of differentiation antigen 20 positive (CD20+) B-cell non-Hodgkin's lymphomas (tissue diagnostic procedures must be performed within 6 months of study entry and with biopsy material available for review):

  * follicular lymphoma (NCI CTCAE grade 1 or 2)
  * immunoplasmacytoma/immunocytoma (Waldenstrom's macroglobulinemia)
  * splenic marginal zone B-cell lymphoma
  * extra-nodal marginal zone lymphoma of mucosa-associated lymphoid tumor (MALT) type
  * nodal marginal zone B-cell lymphoma
  * mantle cell lymphoma
* Meets one of the following need-for-treatment criteria (with the exception of mantle cell lymphoma for which treatment is indicated):

  * presence of at least one of the following B-symptoms:

    1. fever (>38ºC) of unclear etiology
    2. night sweats
    3. weight loss of greater than 10% within the prior 6 months
  * large tumor mass (bulky disease)
  * presence of lymphoma-related complications, including narrowing of ureters or bile ducts, tumor-related compression of a vital organ, lymphoma-induced pain, cytopenias related to lymphoma/leukemia, splenomegaly, pleural effusions, or ascites
  * hyperviscosity syndrome due to monoclonal gammopathy
* CD20+ B cells in lymph node biopsy or other lymphoma pathology specimen.
* No prior treatment (patients on "watch and wait" may enter the study if a recent biopsy [obtained within the last 6 months] is available)
* Adequate hematologic function (unless abnormalities related to lymphoma infiltration of the bone marrow or hypersplenism due to lymphoma) as follows:

  * hemoglobin of >= 10.0 g/dL
  * absolute neutrophil count (ANC) >=1.5*10^9/L
  * platelet count >=100*10^9/L
* Bidimensionally measurable disease (field not previously radiated)
* Able to provide written informed consent
* Eastern Cooperative Oncology Group (ECOG) Performance Status <=2
* Estimated life expectancy >=6 months
* Serum creatinine of <=2.0 mg/dL or creatinine clearance >=50 mL/min
* Alanine aminotransferase (ALT) and aspartate transaminase (AST) ≤2.5*upper limit of normal (ULN), and alkaline phosphatase and total bilirubin within normal limits
* Left ventricular ejection fraction (LVEF) >= 50% by multiple gated acquisition scan (MUGA) or cardiac echocardiogram (ECHO), prior for any patient to be treated with R-CHOP
* A medically accepted method of contraception to be used by women of childbearing potential (not surgically sterile or at least 12 months naturally postmenopausal)
* Men capable of producing offspring and not surgically sterile must practice abstinence or use a barrier method of birth control.

Key Exclusion Criteria:

* Chronic lymphocytic leukemia, small lymphocytic lymphoma (SLL), or grade 3 follicular lymphoma
* Transformed disease (bone marrow blasts are permitted; however, transformed disease indicating leukemic involvement is not permitted)
* Central nervous system (CNS) lymphomatous involvement or leptomeningeal lymphoma
* Prior radiation for NHL, except for a single course of locally delimited radiation therapy with a radiation field not exceeding 2 adjacent lymph node regions
* Active malignancy, other than NHL, within the past 3 years except for localized prostate cancer treated with hormone therapy, cervical carcinoma in situ, breast cancer in situ, or non-melanoma skin cancer following definitive treatment
* New York Heart Association (NYHA) Class III or IV heart failure, arrhythmias or unstable angina, electrocardiograph (ECG) evidence of active ischemia or active conduction system abnormalities, or myocardial infarction within the last 6 months (prior to study entry, ECG abnormalities at screening must be documented by the investigator as not medically relevant)
* Known human immunodeficiency virus (HIV) positivity
* Active hepatitis B or hepatitis C infection (hepatitis B surface antigen testing required)
* Women who are pregnant or lactating
* Corticosteroids for treatment of lymphoma within 28 days of study entry Chronically administered low-dose corticosteroids (e.g., prednisone ≤20 mg/day) for indications other than lymphoma or lymphoma-related complications are permitted
* Any serious uncontrolled, medical or psychological disorder that would impair the ability of the patient to receive therapy
* Any condition which places the patient at unacceptable risk or confounds the ability of the investigators to interpret study data
* Any other investigational agent within 28 days of study entry
* Known hypersensitivity to bendamustine, mannitol, or other study-related drugs
* Ann Arbor stage I disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 447 (Actual)
Dates: Start 2009-04-30; Primary Completion 2012-03-31 (Actual); Study Completion 2012-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor's Medical Expert, Study Director — Cephalon
Locations (128):
- United States (79):
  - Teva Investigational Site 165, Tucson, Arizona
  - Teva Investigational Site 167, Little Rock, Arkansas
  - Teva Investigational Site 11, Corona, California
  - Teva Investigational Site 21, Fountain Valley, California
  - Teva Investigational Site 52, Fountain Valley, California
  - Teva Investigational Site 64, Fullerton, California
  - Teva Investigational Site 40, Los Angeles, California
  - Teva Investigational Site 53, Los Angeles, California
  - Teva Investigational Site 57, San Diego, California
  - Teva Investigational Site 15, Aurora, Colorado
  - Teva Investigational Site 155, Denver, Colorado
  - Teva Investigational Site 5, Fort Collins, Colorado
  - Teva Investigational Site 70, New Britain, Connecticut
  - Teva Investigational Site 37, Norwalk, Connecticut
  - Teva Investigational Site 67, Southington, Connecticut
  - Teva Investigational Site 58, Fort Myers, Florida
  - Teva Investigational Site 38, Hollywood, Florida
  - Teva Investigational Site 23, Jacksonville, Florida
  - Teva Investigational Site 65, Lake Worth, Florida
  - Teva Investigational Site 156, Miami, Florida
  - Teva Investigational Site 160, Orlando, Florida
  - Teva Investigational Site 68, Orlando, Florida
  - Teva Investigational Site 72, Augusta, Georgia
  - Teva Investigational Site 50, Columbus, Georgia
  - Teva Investigational Site 73, Macon, Georgia
  - Teva Investigational Site 49, Centralia, Illinois
  - Teva Investigational Site 48, Chicago, Illinois
  - Teva Investigational Site 9, Chicago, Illinois
  - Teva Investigational Site 14, Normal, Illinois
  - Teva Investigational Site 24, Beech Grove, Indiana
  - Teva Investigational Site 152, Indianapolis, Indiana
  - Teva Investigational Site 31, Iowa City, Iowa
  - Teva Investigational Site 63, Waterloo, Iowa
  - Teva Investigational Site 47, Wichita, Kansas
  - Teva Investigational Site 33, Lexington, Kentucky
  - Teva Investigational Site 19, Shreveport, Louisiana
  - Teva Investigational Site 43, Augusta, Maine
  - Teva Investigational Site 74, Lowell, Massachusetts
  - Teva Investigational Site 22, Duluth, Minnesota
  - Teva Investigational Site 4, Saint Louis Park, Minnesota
  - Teva Investigational Site 162, Columbia, Missouri
  - Teva Investigational Site 157, Kansas City, Missouri
  - Teva Investigational Site 29, Morristown, New Jersey
  - Teva Investigational Site 46, Albuquerque, New Mexico
  - Teva Investigational Site 8, Rochester, New York
  - Teva Investigational Site 10, Syracuse, New York
  - Teva Investigational Site 17, Charlotte, North Carolina
  - Teva Investigational Site 151, Durham, North Carolina
  - Teva Investigational Site 39, Fargo, North Dakota
  - Teva Investigational Site 34, Cincinnati, Ohio
  - Teva Investigational Site 60, Cincinnati, Ohio
  - Teva Investigational Site 28, Cleveland, Ohio
  - Teva Investigational Site 153, Springfield, Oregon
  - Teva Investigational Site 59, Bethlehem, Pennsylvania
  - Teva Investigational Site 44, Danville, Pennsylvania
  - Teva Investigational Site 3, Philadelphia, Pennsylvania
  - Teva Investigational Site 13, Pittsburgh, Pennsylvania
  - Teva Investigational Site 7, Pottstown, Pennsylvania
  - Teva Investigational Site 25, Charleston, South Carolina
  - Teva Investigational Site 71, Columbia, South Carolina
  - Teva Investigational Site 56, Chattanooga, Tennessee
  - Teva Investigational Site 30, Nashville, Tennessee
  - Teva Investigational Site 154, Arlington, Texas
  - Teva Investigational Site 158, Arlington, Texas
  - Teva Investigational Site 6, El Paso, Texas
  - Teva Investigational Site 161, Fort Worth, Texas
  - Teva Investigational Site 159, San Antonio, Texas
  - Teva Investigational Site 166, Sugar Land, Texas
  - Teva Investigational Site 2, Salt Lake City, Utah
  - Teva Investigational Site 18, Abingdon, Virginia
  - Teva Investigational Site 35, Charlottesville, Virginia
  - Teva Investigational Site 164, Norfolk, Virginia
  - Teva Investigational Site 54, Richmond, Virginia
  - Teva Investigational Site 42, Seattle, Washington
  - Teva Investigational Site 150, Spokane, Washington
  - Teva Investigational Site 163, Vancouver, Washington
  - Teva Investigational Site 66, Morgantown, West Virginia
  - Teva Investigational Site 41, Madison, Wisconsin
  - Teva Investigational Site 62, Wausau, Wisconsin
- Australia (17):
  - Teva Investigational Site 315, Perth, Western Australia
  - Teva Investigational Site 305, Concord
  - Teva Investigational Site 317, Douglas
  - Teva Investigational Site 308, East Melbourne
  - Teva Investigational Site 310, Fitzroy
  - Teva Investigational Site 311, Fitzroy
  - Teva Investigational Site 301, Garran
  - Teva Investigational Site 316, Geelong
  - Teva Investigational Site 304, Hobart
  - Teva Investigational Site 312, Kurralta Park
  - Teva Investigational Site 307, Melbourne
  - Teva Investigational Site 318, Parkville
  - Teva Investigational Site 300, South Brisbane
  - Teva Investigational Site 303, Westmead
  - Teva Investigational Site 314, Wodonga
  - Teva Investigational Site 313, Woodville
  - Teva Investigational Site 309, Woolloongabba
- Brazil (11):
  - Teva Investigational Site 503, Barretos
  - Teva Investigational Site 504, Brasília
  - Teva Investigational Site 506, Curitiba
  - Teva Investigational Site 505, Goiânia
  - Teva Investigational Site 502, Jaú
  - Teva Investigational Site 509, Lajeado
  - Teva Investigational Site 507, Porto Alegre
  - Teva Investigational Site 508, Porto Alegre
  - Teva Investigational Site 511, Rio de Janeiro
  - Teva Investigational Site 500, Santo André
  - Teva Investigational Site 501, São Paulo
- Canada (6):
  - Teva Investigational Site 202, Barrie
  - Teva Investigational Site 206, Calgary
  - Teva Investigational Site 200, Halifax
  - Teva Investigational Site 201, Ottawa
  - Teva Investigational Site 203, Vancouver
  - Teva Investigational Site 204, Winnipeg
- Mexico (4):
  - Teva Investigational Site 602, Aguascalientes
  - Teva Investigational Site 603, Hermosillo
  - Teva Investigational Site 600, Monterrey
  - Teva Investigational Site 601, Monterrey
- New Zealand (6):
  - Teva Investigational Site 401, Auckland
  - Teva Investigational Site 405, Auckland
  - Teva Investigational Site 400, Christchurch
  - Teva Investigational Site 402, Newtown
  - Teva Investigational Site 404, Palmerston North
  - Teva Investigational Site 403, Takapuna
- Peru (5):
  - Teva Investigational Site 700, Lima
  - Teva Investigational Site 701, Lima
  - Teva Investigational Site 704, Lima
  - Teva Investigational Site 702, Miraflores
  - Teva Investigational Site 703, Miraflores

REFERENCES:
- [Result] Flinn IW, van der Jagt R, Kahl BS, Wood P, Hawkins TE, Macdonald D, Hertzberg M, Kwan YL, Simpson D, Craig M, Kolibaba K, Issa S, Clementi R, Hallman DM, Munteanu M, Chen L, Burke JM. Randomized trial of bendamustine-rituximab or R-CHOP/R-CVP in first-line treatment of indolent NHL or MCL: the BRIGHT study. Blood. 2014 May 8;123(19):2944-52. doi: 10.1182/blood-2013-11-531327. Epub 2014 Mar 3. PMID 24591201
- [Derived] Flinn IW, van der Jagt R, Kahl B, Wood P, Hawkins T, MacDonald D, Simpson D, Kolibaba K, Issa S, Chang J, Trotman J, Hallman D, Chen L, Burke JM. First-Line Treatment of Patients With Indolent Non-Hodgkin Lymphoma or Mantle-Cell Lymphoma With Bendamustine Plus Rituximab Versus R-CHOP or R-CVP: Results of the BRIGHT 5-Year Follow-Up Study. J Clin Oncol. 2019 Apr 20;37(12):984-991. doi: 10.1200/JCO.18.00605. Epub 2019 Feb 27. PMID 30811293
- [Derived] Burke JM, van der Jagt RH, Kahl BS, Wood P, Hawkins TE, MacDonald D, Hertzberg M, Simpson D, Craig M, Kolibaba K, Issa S, Munteanu M, Victor TW, Flinn IW. Differences in Quality of Life Between Bendamustine-Rituximab and R-CHOP/R-CVP in Patients With Previously Untreated Advanced Indolent Non-Hodgkin Lymphoma or Mantle Cell Lymphoma. Clin Lymphoma Myeloma Leuk. 2016 Apr;16(4):182-190.e1. doi: 10.1016/j.clml.2016.01.001. Epub 2016 Jan 15. PMID 26875824

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 568 participants were screened, and 121 were not randomized (2 due to adverse event, 14 withdrew consent, 68 did not meet inclusion criteria, 23 met exclusion criteria, and 14 for other reasons).
Period: Treatment Period
Arm/Group | Bendamustine and Rituximab (BR) | R-CHOP/R-CVP
Started | 224 | 223
Completed | 199 | 196
Not Completed | 25 | 27
Not completed — Death | 2 | 1
Not completed — Adverse Event | 10 | 3
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Disease Progression | 1 | 2
Not completed — Started New Treatment Regimen | 2 | 5
Not completed — Other | 4 | 4
Not completed — Randomized but Not Treated | 3 | 8
Period: Long-Term Follow-up Period
Arm/Group | Bendamustine and Rituximab (BR) | R-CHOP/R-CVP
Started | 210 | 209
Completed | 157 | 154
Not Completed | 53 | 55
Not completed — Withdrawal by Subject | 12 | 19
Not completed — Lost to Follow-up | 8 | 9
Not completed — Death | 26 | 18
Not completed — Other | 7 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bendamustine and Rituximab (BR) | R-CHOP/R-CVP | Total
Number analyzed (Participants) | 224 | 223 | 447
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (11.37) | 58.2 (12.11) | 59.1 (11.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 91 | 179
  Male | 136 | 132 | 268
European Cooperative Oncology Group Performance Status [Number; unit: participants] — ECOG criteria: 0: Fully active. 1: Ambulatory, carry out work of a light or sedentary nature. 2: Ambulatory, capable of all selfcare. 3: Capable of limited selfcare, confined to bed or chair more than 50% of waking hours. 4: Completely disabled, no selfcare, totally confined to bed or chair. 5: Dead. 1 participant in the R-CHOP/R-CVP treatment group did not have an assessment at baseline.
  participants
    0 | 144 | 143 | 287
    1 | 70 | 69 | 139
    2 | 9 | 10 | 19
    3 | 1 | 0 | 1
    4 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] — one participant in the R-CHOP/R-CVP group did not a a weight measurement at baseline
  kg | 81.9 (18.48) | 82.4 (17.93) | 82.1 (18.19)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Response (CR) at End of Treatment Period
Description: CR=complete disappearance of all detectable clinical evidence of disease and disease-related symptoms, if present pretherapy; protocol-specified positron emission tomography (PET) scan assessment criteria; (if the spleen and/or liver were enlarged on the basis of physical examination and/or anatomic imaging before treatment) the liver and/or spleen were considered normal size on physical examination and by anatomic imaging after therapy, with disappearance of all nodules related to lymphoma; (if the bone marrow was involved by lymphoma before treatment) the infiltrate must have cleared on subsequent bone marrow biopsies.
Time Frame: 6 to 8 21 or 28-day cycles (18-32 weeks)
Population: Evaluable Analysis Set: treated participants with a baseline and >=1 post-baseline response evaluation (based on computed tomography/magnetic resonance imaging [CT/MRI] or positron emission tomography [PET] and clinical data), or who discontinued treatment due to progressive disease and had no major protocol violations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bendamustine and Rituximab (BR) | R-CHOP/R-CVP
Number analyzed (Participants) | 213 | 206
percentage of participants | 31 [25.3 to 38.2] | 25 [19.5 to 31.7]

2. Secondary Outcome: Percentage of Participants With Overall Response at End of Treatment Period
Description: Overall Response=participants with Complete Remission (CR) + those with Partial Remission (PR). CR=see Outcome Measure 1 for details. PR= at least a 50% decrease in the sum of the product of the greatest diameters (SPD) of up to 6 of the largest dominant nodes/masses; at least a 50% decrease in the SPD of hepatic and splenic nodules in their greatest transverse diameter; no increase in the size of the liver, spleen, and other nodes; no measurable disease in organs other than the liver or spleen; no new sites of disease; protocol-specified PET scan and bone marrow criteria.
Time Frame: 6 to 8 21 or 28-day cycles (18-32 weeks)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bendamustine and Rituximab (BR) | R-CHOP/R-CVP
Number analyzed (Participants) | 213 | 206
percentage of participants | 97 [93.3 to 98.7] | 91 [86.0 to 94.4]

3. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Deaths and Discontinuations Due to AEs at End of Treatment Period
Description: AE=any untoward medical occurrence that develops or worsens in severity after dispensation of the study drug and does not necessarily have a causal relationship to the study drug. An AE can, therefore, be any unfavorable and unintended physical sign, symptom, or laboratory parameter that develops or worsens in severity during the course of the study, or significant worsening of the disease under study (or any concurrent disease), whether or not considered related to the study drug. AEs were graded as 1 (mild), 2 (moderate), 3 (severe), 4 (life-threatening), 5 (death). SAE=an adverse event occurring at any dose that results in: death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant disability/incapacity (a substantial disruption of one's ability to conduct normal life functions), a congenital anomaly/birth defect, or other important medical event.
Time Frame: 32 weeks
Population: Safety Analysis Set: all participants randomly assigned to a treatment group who received 1 or more doses of any component of any study drug regimen.
Measure: Number; unit: participants
Arm/Group | Bendamustine and Rituximab (BR) | R-CHOP/R-CVP
Number analyzed (Participants) | 221 | 215
participants
  Any AE | 221 | 213
  Severe AEs (grades 3, 4, 5) | 130 | 127
  Treatment-related AEs | 209 | NA — AE relationship was not assessed (not collected) for participants in the R-CHOP/R-CVP treatment group because it was open label and the events associated with R-CHOP/R-CVP arm were known due to being standard treatment for many countries.
  Deaths | 12 | 9
  SAEs | 60 | 49
  Withdrawn due to AEs | 10 | 3

4. Secondary Outcome: Worst Overall Common Terminology Criteria for Adverse Events (CTCAE) Grades for Serum Chemistry Laboratory Test Results
Description: Clinical laboratory data were graded according to National Cancer Institute's (NCI) CTCAE version 3, and graded as 1 (mild), 2 (moderate), 3 (severe), 4 (life-threatening), 5 (death). The table presents the worst CTCAE grades for serum chemistry test results experienced by participants overall (i.e., the worst post-baseline grade value for each participant and laboratory test across all cycles).
Time Frame: 32 weeks (conducted at screening, Day 1 of each cycle, and end-of-treatment visit)
Population: Safety Analysis Set: all participants randomly assigned to a treatment group who received 1 or more doses of any component of any study drug regimen and who had a post-baseline assessment.
Measure: Number; unit: participants
Arm/Group | Bendamustine and Rituximab (BR) | R-CHOP/R-CVP
Number analyzed (Participants) | 221 | 215
participants
  Albumin: Grade 1 | 33 | 44
  Albumin: Grade 2 | 14 | 13
  Albumin: Grade 3 | 3 | 0
  Albumin: Grade 4 | 0 | 0
  Albumin: Grades 1-4 | 50 | 57
  Alkaline Phosphatase: Grade 1 | 41 | 25
  Alkaline Phosphatase: Grade 2 | 1 | 3
  Alkaline Phosphatase: Grade 3 | 0 | 0
  Alkaline Phosphatase: Grade 4 | 0 | 0
  Alkaline Phosphatase: Grades 1-4 | 42 | 28
  Creatinine: Grade 1 | 19 | 25
  Creatinine: Grade 2 | 3 | 1
  Creatinine: Grade 3 | 1 | 0
  Creatinine: Grade 4 | 0 | 0
  Creatinine: Grades 1-4 | 23 | 26
  Gamma-glutamyl transferase: Grade 1 | 31 | 37
  Gamma-glutamyl transferase: Grade 2 | 18 | 10
  Gamma-glutamyl transferase: Grade 3 | 3 | 6
  Gamma-glutamyl transferase: Grade 4 | 0 | 0
  Gamma-glutamyl transferase: Grades 1-4 | 52 | 53
  Hypercalcemia: Grade 1 | 6 | 6
  Hypercalcemia: Grade 2 | 0 | 0
  Hypercalcemia: Grade 3 | 1 | 0
  Hypercalcemia: Grade 4 | 0 | 0
  Hypercalcemia: Grades 1-4 | 7 | 6
  Hyperglycemia: Grade 1 | 94 | 74
  Hyperglycemia: Grade 2 | 20 | 34
  Hyperglycemia: Grade 3 | 15 | 15
  Hyperglycemia: Grade 4 | 0 | 1
  Hyperglycemia: Grades 1-4 | 129 | 124
  Hyperkalemia: Grade 1 | 7 | 8
  Hyperkalemia: Grade 2 | 3 | 1
  Hyperkalemia: Grade 3 | 1 | 0
  Hyperkalemia: Grade 4 | 0 | 0
  Hyperkalemia: Grades 1-4 | 11 | 9
  Hypernatremia: Grade 1 | 8 | 10
  Hypernatremia: Grade 2 | 0 | 0
  Hypernatremia: Grade 3 | 0 | 0
  Hypernatremia: Grade 4 | 0 | 0
  Hypernatremia: Grades 1-4 | 8 | 10
  Hypocalcemia: Grade 1 | 36 | 28
  Hypocalcemia: Grade 2 | 8 | 6
  Hypocalcemia: Grade 3 | 1 | 0
  Hypocalcemia: Grade 4 | 3 | 0
  Hypocalcemia: Grades 1-4 | 48 | 34
  Hypoglycemia: Grade 1 | 15 | 10
  Hypoglycemia: Grade 2 | 1 | 0
  Hypoglycemia: Grade 3 | 0 | 0
  Hypoglycemia: Grade 4 | 0 | 0
  Hypoglycemia: Grades 1-4 | 16 | 10
  Hypokalemia: Grade 1 | 18 | 16
  Hypokalemia: Grade 2 | 0 | 0
  Hypokalemia: Grade 3 | 0 | 1
  Hypokalemia: Grade 4 | 0 | 0
  Hypokalemia: Grades 1-4 | 18 | 17
  Hyponatremia: Grade 1 | 40 | 28
  Hyponatremia: Grade 2 | 0 | 0
  Hyponatremia: Grade 3 | 0 | 5
  Hyponatremia: Grade 4 | 0 | 0
  Hyponatremia: Grades 1-4 | 40 | 33
  Magnesium: Grade 1 | 46 | 44
  Magnesium: Grade 2 | 0 | 1
  Magnesium: Grade 3 | 0 | 1
  Magnesium: Grade 4 | 0 | 0
  Magnesium: Grades 1-4 | 46 | 46
  Phosphorus: Grade 1 | 7 | 5
  Phosphorus: Grade 2 | 25 | 22
  Phosphorus: Grade 3 | 3 | 3
  Phosphorus: Grade 4 | 0 | 1
  Phosphorus: Grades 1-4 | 35 | 31
  Aspartate Aminotransferase: Grade 1 | 42 | 32
  Aspartate Aminotransferase: Grade 2 | 2 | 2
  Aspartate Aminotransferase: Grade 3 | 1 | 1
  Aspartate Aminotransferase: Grade 4 | 0 | 0
  Aspartate Aminotransferase: Grades 1-4 | 45 | 35
  Alanine Aminotransferase: Grade 1 | 46 | 38
  Alanine Aminotransferase: Grade 2 | 6 | 3
  Alanine Aminotransferase: Grade 3 | 2 | 1
  Alanine Aminotransferase: Grade 4 | 0 | 0
  Alanine Aminotransferase: Grades 1-4 | 54 | 42
  Total Bilirubin: Grade 1 | 14 | 7
  Total Bilirubin: Grade 2 | 1 | 0
  Total Bilirubin: Grade 3 | 0 | 0
  Total Bilirubin: Grade 4 | 0 | 0
  Total Bilirubin: Grades 1-4 | 15 | 7
  Uric Acid: Grade 1 | 41 | 42
  Uric Acid: Grade 2 | 0 | 0
  Uric Acid: Grade 3 | 0 | 0
  Uric Acid: Grade 4 | 1 | 0
  Uric Acid: Grades 1-4 | 42 | 42

5. Secondary Outcome: Worst Overall CTCAE Grade for Hematology Laboratory Test Results
Description: Hematology test data were graded according to National Cancer Institute's (NCI) CTCAE version 3, and graded as 1 (mild), 2 (moderate), 3 (severe), 4 (life-threatening), 5 (death). The table presents the worst CTCAE grades for hematology test results experienced by participants overall (i.e., the worst post-baseline grade value for each participant and hematology test across all cycles).
Time Frame: 32 weeks (conducted at screening, Day 1 of each cycle, weekly during treatment, and at the end-of-treatment visit)
Population: Safety Analysis Set: all participants randomly assigned to a treatment group who received 1 or more doses of any component of any study drug regimen and who had an assessment.
Measure: Number; unit: participants
Arm/Group | Bendamustine and Rituximab (BR) | R-CHOP/R-CVP
Number analyzed (Participants) | 221 | 215
participants
  Absolute Neutrophil Count: Grade 1 | 22 | 14
  Absolute Neutrophil Count: Grade 2 | 51 | 20
  Absolute Neutrophil Count: Grade 3 | 48 | 47
  Absolute Neutrophil Count: Grade 4 | 50 | 104
  Absolute Neutrophil Count: Grades 1-4 | 171 | 185
  Hemoglobin: Grade 1 | 129 | 129
  Hemoglobin: Grade 2 | 42 | 51
  Hemoglobin: Grade 3 | 5 | 7
  Hemoglobin: Grade 4 | 1 | 2
  Hemoglobin: Grades 1-4 | 177 | 189
  Lymphocytes Absolute: Grade 1 | 1 | 6
  Lymphocytes Absolute: Grade 2 | 5 | 55
  Lymphocytes Absolute: Grade 3 | 54 | 55
  Lymphocytes Absolute: Grade 4 | 83 | 9
  Lymphocytes Absolute: Grades 1-4 | 143 | 125
  Platelets: Grade 1 | 106 | 72
  Platelets: Grade 2 | 14 | 14
  Platelets: Grade 3 | 9 | 7
  Platelets: Grade 4 | 7 | 8
  Platelets: Grades 1-4 | 136 | 101
  White Blood Cells: Grade 1 | 41 | 22
  White Blood Cells: Grade 2 | 79 | 49
  White Blood Cells: Grade 3 | 65 | 89
  White Blood Cells: Grade 4 | 19 | 27
  White Blood Cells: Grades 1-4 | 204 | 187

6. Secondary Outcome: Clinically Significant Abnormal Vital Signs
Time Frame: 32 weeks (conducted at screening, Day 1 of each cycle, and end-of-treatment visit)
Population: Safety Analysis Set: all participants randomly assigned to a treatment group who received 1 or more doses of any component of any study drug regimen and had baseline and post-baseline values.
Measure: Number; unit: participants
Arm/Group | Bendamustine and Rituximab (BR) | R-CHOP/R-CVP
Number analyzed (Participants) | 220 | 212
participants
  Heart Rate >=120 and ↑ >=15 bpm | 0 | 1
  Heart Rate <=50 and ↓ >=15 bpm | 2 | 2
  Systolic Blood Pressure(BP) >=180 and ↑ >=20 mm Hg | 2 | 2
  Systolic BP <=90 and ↓ >=20 mm Hg | 6 | 2
  Diastolic BP >=105 and ↑ from Baseline >=15 mm Hg | 1 | 2
  Diastolic BP <=50 and ↓ from Baseline >=15 mm Hg | 2 | 2

7. Secondary Outcome: Potentially Clinically Significant Abnormal Weight
Description: Participants were weighed at Baseline and at Endpoint (Week 32); those participants with an increase or decrease of >=10% were considered potentially clinically significant.
Time Frame: Baseline, Week 32
Population: Safety Analysis Set: all participants randomly assigned to a treatment group who received 1 or more doses of any component of any study drug regimen with a baseline and post-baseline weight.
Measure: Number; unit: participants
Arm/Group | Bendamustine and Rituximab (BR) | R-CHOP/R-CVP
Number analyzed (Participants) | 220 | 212
participants
  Increase >=10% | 8 | 5
  Decrease >=10% | 18 | 8

8. Secondary Outcome: Eastern Cooperative Oncology Group (ECOG) Performance Status at the End of Treatment Period
Description: Participants' ECOG Performance Status was evaluated at the end of treatment as improved, stayed the same, or worsened from baseline (see Baseline Characteristics for ECOG Performance Status).
Time Frame: Week 32
Population: Safety Analysis Set: all participants randomly assigned to a treatment group who received 1 or more doses of any component of any study drug regimen and with baseline and post-baseline values.
Measure: Number; unit: participants
Groups:
- Bendamustine/Rituximab: bendamustine at 90 mg/m2 iv on days 1 and 2 and rituximab at 375 mg/m2 iv infusion on day 1
- R-CHOP/R-CVP: R-CHOP, consisting of rituximab at 375 mg/m2 iv on day 1, vincristine at 1.4 mg /m2 (up to a maximum dose of 2 mg iv) by iv on day 1, prednisone at 100 mg orally on days 1 to 5 of a 21-day cycle, doxorubicin at 50 mg/m2 by iv over 3-5 minutes on day 1, cyclophosphamide iv at 750 mg/m2 on day 1.
  R-CVP consisting of rituximab at 375 mg/m2 iv on day 1, vincristine at 1.4 mg /m2 (up to a maximum dose of 2 mg iv) by iv on day 1, prednisone at 100 mg orally on days 1 to 5 of a 21-day cycle, only 1 of the following doses of cyclophosphamide throughout the study: cyclophosphamide at 750 mg/m2 iv on day 1 or cyclophosphamide at 1000 mg/m2 iv on day 1.
Arm/Group | Bendamustine/Rituximab | R-CHOP/R-CVP
Number analyzed (Participants) | 219 | 211
participants
  Improved | 32 | 28
  Stayed the Same | 153 | 141
  Worsened | 34 | 42

9. Secondary Outcome: Therapeutic Classification of Prior Medications
Time Frame: prior to start of treatment
Population: Safety Analysis Set: all participants randomly assigned to a treatment group
Measure: Number; unit: participants
Arm/Group | Bendamustine and Rituximab (BR) | R-CHOP/R-CVP
Number analyzed (Participants) | 224 | 223
participants
  Psycholeptics | 57 | 59
  Sex Hormones and Modulators of the Genital System | 11 | 12
  Stomatological Preparations | 0 | 0
  Throat Preparations | 0 | 0
  Thyroid Therapy | 16 | 17
  Topical Products for Join and Muscular Pain | 1 | 0
  Unspecified Herbal | 10 | 10
  Urologicals | 20 | 11
  Vaccines | 2 | 7
  Vasoprotectives | 0 | 0
  Vitamins | 70 | 61

10. Secondary Outcome: Therapeutic Classification of Concomitant Medications
Time Frame: 32 weeks
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Bendamustine and Rituximab (BR) | R-CHOP/R-CVP
Number analyzed (Participants) | 221 | 215
participants
  Psycholeptics | 69 | 74
  Sex Hormones and Modulators of the Genital System | 6 | 4
  Stomatological Preparations | 23 | 29
  Throat Preparations | 3 | 2
  Thyroid Therapy | 3 | 1
  Topical Preparations for Join and Muscular Pain | 1 | 2
  Unspecified Herbal | 3 | 5
  Urologicals | 5 | 4
  Vaccines | 11 | 11
  Vasoprotectives | 1 | 8
  Vitamins | 16 | 21

11. Secondary Outcome: Change From Baseline to End of Treatment in the Global Health Status Score of the European Organization for Research and Treatment of Cancer (EORTC) 30-item Core Quality of Life Questionnaire (QLQ-C30)
Description: EORTC QLQ-C30 is a 30-item questionnaire to assess the overall quality of life in cancer patients. EORTC QLQ-C30 includes functional scales (physical, role, cognitive, emotional, and social), global health status, symptom scales (fatigue, pain, nausea/vomiting), and other (dyspnoea, appetite loss, insomnia, constipation/diarrhea, and financial difficulties). This outcome reports the global health status on a scale of 0-100 with a high score for the global health status/QOL represents a high quality of life.
Time Frame: Day 1 (prior to treatment), 32 weeks
Population: The set of randomized participants (intent-to-treat) consisting of all patients randomly assigned to treatment, and who had data at both timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bendamustine and Rituximab (BR) | R-CHOP/R-CVP
Number analyzed (Participants) | 211 | 207
units on a scale | 3.6 (24.60) | -5.1 (24.50)
Statistical Analysis 1: Comparison: Bendamustine and Rituximab (BR) vs R-CHOP/R-CVP; The hypothesis of interest is superiority of BR over standard treatment; Test type: Superiority or Other; p = 0.0005, ANCOVA — P-value for the treatment comparison is from an analysis of covariance (ANCOVA) with treatment group, region, preassigned standard treatment, and lymphoma type as factors and baseline value as the covariate

12. Secondary Outcome: Participants With Disease Progression, Relapse or Death At the End of the Treatment Period or the Long-Term Follow-up Period
Description: Relapsed disease (after CR) and progressive disease (PD) (after PR or SD):
  * Lymph nodes were considered abnormal if the long axis was greater than 1.5 cm. Lymph nodes with a long axis of 1.1 to 1.5 cm were considered abnormal if its short axis was greater than 1.0 cm.
  * In patients with no prior history of pulmonary lymphoma, new lung nodules identified by CT require histologic confirmation.
  * >= 50% increase from nadir in sum of the products of the greatest diameters (SPD) of any previously involved nodes, or in a single involved node, or the size of other lesions (eg, splenic or hepatic nodules). To be considered progressive disease, a lymph node with a diameter of the short axis of less than 1.0 cm must have increased by 2: 50% and to a size of 1.5 cm by 1.5 cm, or more than 1.5 cm in the long axis
  * other conditions as specified in the protocol
Time Frame: Treatment Period: 18-32 weeks Long-Term Follow-up Period: up to 5 years after the Treatment Period
Population: Randomized patients: the set of randomized patients (intent-to-treat) consists of all patients randomly assigned to treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Bendamustine and Rituximab (BR) | R-CHOP/R-CVP
Number analyzed (Participants) | 224 | 223
Participants | 36 | 30
Statistical Analysis 1: Comparison: Bendamustine and Rituximab (BR) vs R-CHOP/R-CVP; Test type: Superiority; p = 0.9677, Log Rank; Stratified log-rank test by preassigned standard treatment and lymphoma type; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.58 to 1.68] — BR/RCHOP-RCVP

13. Secondary Outcome: Kaplan-Meier Estimate for Progression-free Survival (PFS)
Description: PFS was defined as the time from randomization to disease progression or relapse, or death from any cause, whichever occurred first.
Time Frame: Day 1 up to 5.6 years (Treatment Period + Long-Term Follow-up Period)
Population: Randomized patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bendamustine and Rituximab (BR) | R-CHOP/R-CVP
Number analyzed (Participants) | 224 | 223
months | 31.8 [16.9 to 43.2] | 33.4 [19.3 to 48.7]

14. Secondary Outcome: Kaplan-Meier Estimate for Event-free Survival (EFS)
Description: EFS was defined as the time from randomization to treatment failure, disease progression or relapse, other malignancies, or death from any cause, whichever occurred first.
  Treatment failure was defined as failure to achieve a CR or PR after 6 cycles of treatment. If a patient failed to achieve CR or PR by the time of data analysis or early withdrawal, the treatment failure date was set at 126 days (6 cycles of treatment) after randomization or the new anticancer treatment date, whichever is earlier.
Time Frame: Day 1 up to 5.6 years (Treatment Period + Long-Term Follow-up Period)
Population: Randomized patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bendamustine and Rituximab (BR) | R-CHOP/R-CVP
Number analyzed (Participants) | 224 | 223
months | 31.8 [15.5 to 43.2] | 32.6 [18.1 to 44.7]

15. Secondary Outcome: Kaplan-Meier Estimate for Duration of Response (DOR)
Description: DOR was defined as the time from first response (CR or PR) to disease progression or relapse, or death due to any cause.
Time Frame: Day 1 up to 5.6 years (Treatment Period + Long-Term Follow-up Period)
Population: Randomized patients with complete response (CR) or partial response (PR)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bendamustine and Rituximab (BR) | R-CHOP/R-CVP
Number analyzed (Participants) | 210 | 187
months | 26.5 [12.8 to 42.9] | 32.1 [19.8 to 46.7]

16. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death from any cause.
Time Frame: Day 1 up to 5.6 years (Treatment Period + Long-Term Follow-up Period)
Population: Randomized patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bendamustine and Rituximab (BR) | R-CHOP/R-CVP
Number analyzed (Participants) | 224 | 223
months | 65.0 [64.8 to 65.1] | 64.1 [63.8 to 64.3]

17. Secondary Outcome: Participants Who Died At the End of the Treatment Period or the Long-Term Follow-up Period
Description: Death is due to any cause. Data are broken out by patients who died within 30 days of the last dose of study medications, and those who died greater than 30 days of the last dose of study medications.
Time Frame: Treatment Period: 18-32 weeks Long-Term Follow-up Period: up to 5 years after the Treatment Period
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Bendamustine and Rituximab (BR) | R-CHOP/R-CVP
Number analyzed (Participants) | 224 | 223
Participants
  All Deaths | 40 | 32
  Deaths within 30 days of study treatment | 2 | 1
  Deaths greater than 30 days of study treatment | 38 | 31

ADVERSE EVENTS:
Time Frame: Treatment Period: 32 weeks No adverse event data was collected during the 5-year Long-Term Follow-Up Period
Description: Events are reported for the safety analysis set (participants who received at least 1 dose of study drug).
Groups:
- R-CHOP/CVP: Participants received the standard regimen (R-CHOP or R-CVP) for 6 to 8 21-days cycles.
  R-CHOP: rituximab 375 mg/m^2 IV on Day 1; vincristine 1.4 mg/m^2 (up to 2 mg/m^2 maximum dose) IV on Day 1; doxorubicin 50 mg/m^2 IV Day 1; cyclophosphamide 750 mg/m^2 IV Day 1; prednisone 100 mg oral on Days 1 to 5
  R-CVP: rituximab 375 mg/m^2 IV on Day 1; cyclophosphamide 750 mg/m^2 IV on Day 1 or cyclophosphamide 1000 mg/m^2 IV on Day 1; vincristine 1.4 mg/m^2 (up to 2 mg/m^2 maximum dose) IV on Day 1; prednisone 100 mg oral on Days 1 to 5
Arm/Group | Bendamustine and Rituximab (BR) | R-CHOP/CVP
Serious Adverse Events (participants affected / at risk) | 60/221 | 49/215
Other Adverse Events (participants affected / at risk) | 216/221 | 211/215
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bendamustine and Rituximab (BR) (N=221) | R-CHOP/CVP (N=215)
Aplasia pure red cell (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 (8) | 9 (10)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 4 (6) | 5 (6)
Splenomegaly (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0)
Bundle branch block left (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 1 (2)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Vitreous floaters (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Chills (General disorders) | 1 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 3 (3)
Pyrexia (General disorders) | 5 (6) | 4 (5)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Anaphylactic shock (Immune system disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 4 (4) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Anal infection (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 2 (3) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumocystis jiroveci infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 7 (7) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 1 (2)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 2 (2) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 8 (11) | 4 (4)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dystonia (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bendamustine and Rituximab (BR) (N=221) | R-CHOP/CVP (N=215)
Anaemia (Blood and lymphatic system disorders) | 31 (63) | 29 (69)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 (9) | 11 (12)
Leukopenia (Blood and lymphatic system disorders) | 21 (79) | 22 (88)
Lymphopenia (Blood and lymphatic system disorders) | 14 (104) | 12 (44)
Neutropenia (Blood and lymphatic system disorders) | 76 (251) | 85 (255)
Thrombocytopenia (Blood and lymphatic system disorders) | 29 (67) | 13 (54)
Abdominal pain (Gastrointestinal disorders) | 25 (33) | 27 (31)
Abdominal pain upper (Gastrointestinal disorders) | 11 (11) | 14 (16)
Constipation (Gastrointestinal disorders) | 65 (85) | 90 (121)
Diarrhoea (Gastrointestinal disorders) | 46 (65) | 50 (72)
Dyspepsia (Gastrointestinal disorders) | 23 (23) | 26 (29)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 16 (16) | 17 (18)
Nausea (Gastrointestinal disorders) | 139 (255) | 102 (139)
Stomatitis (Gastrointestinal disorders) | 15 (20) | 14 (17)
Vomiting (Gastrointestinal disorders) | 60 (86) | 28 (35)
Asthenia (General disorders) | 14 (16) | 17 (24)
Chest discomfort (General disorders) | 8 (10) | 13 (14)
Chills (General disorders) | 25 (34) | 11 (14)
Fatigue (General disorders) | 113 (179) | 107 (147)
Mucosal inflammation (General disorders) | 12 (15) | 26 (36)
Oedema peripheral (General disorders) | 19 (23) | 23 (27)
Pain (General disorders) | 14 (15) | 14 (17)
Pyrexia (General disorders) | 37 (45) | 28 (31)
Drug hypersensitivity (Immune system disorders) | 24 (32) | 8 (9)
Nasopharyngitis (Infections and infestations) | 9 (9) | 11 (11)
Sinusitis (Infections and infestations) | 5 (7) | 12 (14)
Upper respiratory tract infection (Infections and infestations) | 22 (26) | 17 (20)
Infusion related reaction (Injury, poisoning and procedural complications) | 52 (115) | 45 (64)
Neutrophil count decreased (Investigations) | 9 (15) | 12 (18)
Weight decreased (Investigations) | 14 (14) | 7 (8)
Decreased appetite (Metabolism and nutrition disorders) | 42 (57) | 26 (26)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (9) | 11 (26)
Arthralgia (Musculoskeletal and connective tissue disorders) | 28 (33) | 32 (46)
Back pain (Musculoskeletal and connective tissue disorders) | 23 (26) | 27 (39)
Bone pain (Musculoskeletal and connective tissue disorders) | 9 (10) | 18 (20)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 (6) | 11 (14)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 12 (12) | 17 (18)
Myalgia (Musculoskeletal and connective tissue disorders) | 13 (15) | 18 (21)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 17 (23) | 18 (20)
Dizziness (Nervous system disorders) | 18 (31) | 21 (29)
Dysgeusia (Nervous system disorders) | 28 (32) | 25 (25)
Headache (Nervous system disorders) | 48 (60) | 45 (68)
Neuropathy peripheral (Nervous system disorders) | 9 (13) | 51 (77)
Paraesthesia (Nervous system disorders) | 7 (8) | 25 (29)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (4) | 20 (24)
Anxiety (Psychiatric disorders) | 17 (18) | 18 (20)
Insomnia (Psychiatric disorders) | 37 (42) | 47 (53)
Cough (Respiratory, thoracic and mediastinal disorders) | 34 (37) | 34 (36)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 (23) | 26 (28)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 18 (20) | 16 (18)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (8) | 74 (83)
Dry skin (Skin and subcutaneous tissue disorders) | 12 (13) | 7 (7)
Night sweats (Skin and subcutaneous tissue disorders) | 7 (7) | 15 (15)
Pruritus (Skin and subcutaneous tissue disorders) | 22 (26) | 10 (10)
Rash (Skin and subcutaneous tissue disorders) | 33 (40) | 17 (20)
Hypotension (Vascular disorders) | 12 (13) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator/Institution must submit proposed publication to Sponsor for review within a prespecified number of days before submission for publication. If Sponsor's review shows that potentially patentable subject matter would be disclosed, publication/public disclosure shall be delayed to enable Sponsor, or Sponsor's designees, to file necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.